CLINICAL TRIAL: NCT05860530
Title: Bioequivalence Study of Two Olaparib Tablets in Patients With Cancers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: QL-YK3-052-001
Record Dates: First submitted 2023-05-08; First posted 2023-05-16 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test-reference (Other): Administration order: The test olaparib tablets for 7 days, then the reference olaparib tablets for 7 days.
  Interventions: Drug: The test olaparib tablet (T); Drug: The reference olaparib tablet (R)
- Reference-test (Other): Administration order: The reference olaparib tablets for 7 days, then the test olaparib tablets for 7 days.
  Interventions: Drug: The test olaparib tablet (T); Drug: The reference olaparib tablet (R)

INTERVENTIONS:
Drug: The test olaparib tablet (T) — The test olaparib tablet (Qilu Pharmaceutical Co., Ltd., Jinan, China) 300mg, every 12 hours
Drug: The reference olaparib tablet (R) — The reference olaparib tablet (Lynparza®; AstraZeneca PLC, Cambridge, England, UK) 300mg, every 12 hours

SUMMARY:
This study aimed to evaluate the pharmacokinetic characteristics and bioequivalence of two olaparib tablets in patients with epithelial ovarian, fallopian tube, or primary peritoneal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Had BMI 18.0 kg/m^2, and weight ≥ 50 kg for male, or ≥ 45 kg for female
* Patients who were on olaparib treatment, had epithelial ovarian, fallopian tube, or primary peritoneal cancer, or were eligible for olaparib treatment judged investigators
* Had ECOG performance status 0-1
* Had life expectancy >12 weeks
* Had Adequate organ function or clinically irrelevant abnormal result
* Agreed to use adequate contraception from 14 days before treatment initiation to 6 months after last dose

Exclusion Criteria:

* Allergic to any component of study drugs
* Had central nervous system metastases (stable and asymptomatic metastases were acceptable)
* Had other malignancy within 5 years
* Had disease affecting swallow or absorption
* Received major surgery within 1 month before study drug administration
* Had major disease
* Had continuous grade 3-4 adverse event
* Had drug abuse
* Had (suspected) pneumonitis
* Participated in other clinical trial of drug or device within 1 month
* Lost or donated blood > 200 mL or received blood transfusion within 1 month
* With average alcohol consumption > 14 units/week or cigarette consumption > 20/day within 1 month
* Positive for human immunodeficiency virus, hepatitis B, C, or syphilis test
* Received strong or moderate CYP3A inducer or inhibitor within 3 half-lives of the drug
* Consumed grape fruit juice, or other food or beverage containing caffeine or xanthine
* For female, pregnant or breastfeeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2021-09-08 (Actual); Study Completion 2021-09-08 (Actual)

PRIMARY OUTCOMES:
Cmax,ss | Day 7
  The maximum plasma drug concentration at steady state
AUC0-τ | 0-12 hours
  The area under the concentration-time curve between two dosings at steady state

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui, China